CLINICAL TRIAL: NCT04735133
Title: The Effect of Surgical Wound Complications Profilactic Negative Pressure Wound Therapy in Patients With High Risk Colorectal Cancer Surgery
Brief Title: The Effect of Wound Problems Wound Dressing in Patients With Colorectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Hatice Yüceler Kaçmaz, Research Sssistant (PhD), TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TDK-2018-8406
Record Dates: First submitted 2021-01-26; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Cancer; Surgery; Surgery--Complications; Surgical Site Infection; Wound Complication
Keywords: colorectal cancer; colorectal surgery; surgical site infection; surgical wound complication; negative pressure wound therapy
MeSH Terms: conditions — Colorectal Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention grpup (Experimental): pNPWT device was placed in the pNPWT group for seven days. The incision area was evaluated during the first seven days, and on the 15th, 21st, and 30th days postoperatively for the presence of hematoma, seroma, wound dehiscence/evisceration, and SSI.
  Interventions: Device: pNBYT
- control group (No Intervention): The wound of the control group was covered with a sterile gauze dressing. After the wound was left closed for 48 hours in the clinical routine, the surgical site was left open, supporting healing. Therefore, the dressing of the control group was removed after 48 hours, and the wound was left open.
  The incision area was evaluated during the first seven days, and on the 15th, 21st, and 30th days postoperatively for the presence of hematoma, seroma, wound dehiscence/evisceration, and SSI.

INTERVENTIONS:
Device: pNBYT — pNPWT device (80mm Hg) was placed in the pNPWT group for seven days The incision area was evaluated during the first seven days, and on the 15th, 21st, and 30th days postoperatively for the presence of hematoma, seroma, wound dehiscence/evisceration, and SSI.
  Arms: intervention grpup

SUMMARY:
This study was conducted as a randomized controlled trial in order to determine the effect of prophylactic negative pressure wound therapy for the prevention of surgical site complications in high-risk colorectal cancer surgery.

Hypothesis: Prophylactic negative pressure wound therapy applied after open colorectal cancer surgery to high-risk patients affects surgical wound complications.

pNBYT group: The study was completed with a total of 50 patients, 24 of intervention group anda 26 of the control group, who met the inclusion criteria at the surgical oncology service of a university hospital.

The data were collected using Patient Identification Form, Surgical Procedure Form, Wound Follow-up Chart and ASEPSİS Wound Scoring System. Ethics committee approval and written informed consent of the individuals was taken in the research.

The data were analyzed in SPSS Statistics 24.0 program using Shapiro Wilk test and Q-Q graphs, Independent Sample t test, Mann Whitney U test, Chi-square, Cochran's Q and Friedman test. The value of p<0.05 was accepted for the statistical significance level. It was determined that the groups were similar in terms of identification and surgical procedure characteristics.

DETAILED DESCRIPTION:
The effects of negative pressure wound treatment applied to high-risk patients after open colorectal cancer surgery on four SWCs, including surgical site infections, hematoma, seroma, and wound dehiscence, were studied. The study started before surgery and lasted up to one month after surgery.

Preoperatively, patients fasted for eight hours before the operation and were required to take a shower with 2% chlorhexidine gluconate at night. The patients who required surgical hair removal were shaved with a clipper in the operating room before the operation. Also, patients received 1g of ampicillin + sulbactam/cefazolin within 60 minutes before the incision.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing open colorectal cancer surgery, clean-contaminated (Class-II) or contaminated (Class-III) wounds, ASA 2, 3, or 4, and fulfilling at least one of the following criteria were included:

* 75 years old and above,
* Chronic disease such as Diabetes (DM), Chronic obstructive pulmonary disease (COPD), Heart failure (Ejection fraction ≤ 40%), Preoperative anemia (Hb≤10mg/dl),
* Nutritional problems (BMI 30 kg / m2 and over, malnutrition (NRS 2002 score 3 and over or albumin≤3 mg/dl),
* Regular steroids or anticoagulants,
* Neoadjuvant chemotherapy and radiotherapy.

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
surgical wound complications (SWC) | postoperative 30th day
  surgical site infection, seroma, hematoma, wound dehiscence/evisceration

SECONDARY OUTCOMES:
The ASEPSIS Wound Scoring System | All participants will be followed up 4 times during a month (seven days, 15th, 21st, and 30th days
  is a quantitative scoring method that provides a numerical value regarding the severity of the SSI by using objective criteria based on the appearance of the wound. The wound score is categorized into five stages: 0-10 points are considered satisfactory healing, 11-20 points disturbance of healing, 21-30 points minor wound infection, 31-40 points moderate wound infection, and ≥41 points severe wound infection.
length of stay in the hospital | 30days

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kacmaz HY, Baser M, Sozuer EM. Effect of Prophylactic Negative-Pressure Wound Therapy for High-Risk Wounds in Colorectal Cancer Surgery: A Randomized Controlled Trial. Adv Skin Wound Care. 2022 Nov 1;35(11):597-603. doi: 10.1097/01.ASW.0000874168.60793.10. PMID 36264751